CLINICAL TRIAL: NCT02240693
Title: A Multi-centre, Double-blind, Parallel-group, Randomized Controlled Study to Investigate the Efficacy, Safety and Tolerability of Orally Administered BI 409306 During a 12-week Treatment Period Compared to Placebo in Patients With Alzheimer Disease
Brief Title: Alzheimer Disease Proof of Concept Study With BI 409306 Versus Placebo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1289.5; 2013-005031-24 (EudraCT Number)
Record Dates: First submitted 2014-09-15; First posted 2014-09-16 (Estimated); Results first posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — BI 409306

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- BI 409306 dose 1 (Experimental)
  Interventions: Drug: BI 409306; Drug: Placebo
- BI 409306 dose 2 (Experimental)
  Interventions: Drug: Placebo; Drug: BI 409306
- BI 409306 dose 3 (Experimental)
  Interventions: Drug: BI 409306; Drug: Placebo
- BI 409306 dose 4 (Experimental)
  Interventions: Drug: BI 409306; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 409306
  Arms: BI 409306 dose 1
Drug: Placebo
  Arms: BI 409306 dose 2
Drug: BI 409306
  Arms: BI 409306 dose 2
Drug: Placebo
  Arms: Placebo
Drug: Placebo
  Arms: BI 409306 dose 1
Drug: BI 409306
  Arms: BI 409306 dose 3
Drug: BI 409306
  Arms: BI 409306 dose 4
Drug: Placebo
  Arms: BI 409306 dose 3
Drug: Placebo
  Arms: BI 409306 dose 4

SUMMARY:
The study is designed to compare the effects of 4 different doses of orally administered BI 409306 to placebo in patients with Alzheimers Disease

ELIGIBILITY:
Inclusion criteria:

* Male and female patients with an age of at least 55 years
* Body weight not lower than 50 kgs
* Patients with a confirmed diagnosis of prodromal Alzheimer's Dementia (AD) on neuropsychological testing defined as:

Mini-Mental State Examination (MMSE) score: greater or equal 24 and a global Clinical Dementia Rating (CDR)-score of 0 or 0.5 and

Free and Cued Selective Recall Reminding Test (FCSRT) score:

free recall test: lower or equal 20 (out of 48) and total recall test: lower or equal 42 (out of 48)

Patients who do not reach the required score in FCSRT will additionally perform the Wechsler Memory Visual Paired Associates test. If the Wechsler Memory Visual Paired Associates test shows a cognitive deficit worse than 1 standard deviation to the mean (compared to the reference values of age and educational norms for inclusion), then the patients can be considered to be eligible for the study.

* Confirmation of abnormal markers of AD pathology either via a), or alternatively b) mentioned below:

  1. Presence in cerebrospinal fluid of (samples taken within past 4 months may be eligible,:

     low Aß1-42 concentrations (< 640 pg/mL) and increased total tau concentrations (> 375 pg/ml), or / and low Aß1-42 concentrations (< 640 pg/mL) and increased phospho-tau concentrations (> 52 pg/mL in cerebrospinal fluid), or
  2. Abnormal amyloid deposition in a cerebral Positron Emission Tomography (PET) scan. Scans performed in the past according to the recommendation in the protocol are acceptable
* Patients who have not received prescribed drugs for treatment of AD (including acetyl cholinesterase inhibitors (donepezil, galantamine, rivastigmine, tacrine, phenserine) and Memantine within three months prior to screening
* Patients must have at least 6 years of formal education and fluency in the test language as verbally confirmed by the patient and documented by the study investigator.
* Patients must have given written informed consent in accordance with Good Clinical Practice (GCP) and local legislation prior to any study procedures. All patients must be able to give informed consent personally and have capacity for such consent. An informed consent given by a legal representative will not be accepted.
* Patients must have a reliable study partner (per investigator judgement, for instance a family member, partner, guardian etc.)

Exclusion criteria:

* Mild cognitive impairment with any etiology other than prodromal AD (for example: neurosyphilis, craniocerebral trauma, small vessel disease) based on clinical data and/or current laboratory findings and/or a pre-existing MRI or CT of the brain (CCT). If previous cranial imaging is not available or older than 12 months prior to screening then a CCT or MRI needs to be performed at screening
* Substantial concomitant cerebrovascular disease (defined by a history of a stroke / intracranial haemorrhagia) temporally related to the onset of worsening of cognitive impairment per investigator judgement
* Medical history of cancer (except for basal cell carcinoma) and/or treatment for cancer within the last 5 years
* Medical history or diagnosis of any of symptomatic and unstable/uncontrolled conditions per investigator judgement
* Severe renal impairment defined with a glomerular filtration rate (GFR) < 30ml/min/1.73m2 in the screening central lab report
* Any other psychiatric disorders such as schizophrenia, or mental retardation
* Any suicidal actions in the past 2 years (per investigator judgement i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behaviour)
* Any suicidal ideation of type 4 or 5 in the Columbia Suicide Severity Rating Scale (C-SSRS) in the past 3 months (i.e. active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent)
* Previous participation in investigational drug studies of mild cognitive impairment within three months prior to screening. Having received active treatment in any other study targeting disease modification like Aß immunization and tau therapies. Previous participation in studies with non-prescription medications, vitamins or other nutritional formulations is allowed.
* Significant history of drug dependence or abuse (including alcohol, as defined in Diagnostic and Statistical Manual of Mental Disorders [DSM-V] or in the opinion of the investigator) within the last two years, or a positive urine drug screen for cocaine, heroin, or marijuana.
* Known history of HIV infection
* Any planned surgeries requiring general anaesthesia, or hospitalisation for more than 1 day during the study period
* Pre-menopausal women (last menstruation <= 1 year prior to informed consent) who are nursing or pregnant or are of child-bearing potential and are not practicing an acceptable method of birth control
* For male patients: Men who are able to father a child, unwilling to be abstinent or to use an adequate form of effective contraception for the duration of study participation and for at least 28 days after treatment has ended.
* Use of any investigational drug or procedure for other indications within 3 months or 6 half-lives (whichever is longer) prior to randomization.
* Intake of the following medications within 3 months prior to randomization and intended to be initiated during the duration of the trial:

  1. tricyclic antidepressants,
  2. antidepressants that are monoamine oxidase inhibitors,
  3. neuroleptics with moderate or greater anticholinergic potency (e.g. chlorpromazine, fluphenazine, loxapine, perphenazine, thioridazine),
  4. anticholinergic medications

The following drugs may be given as needed if the total daily dose was stable 8 weeks prior to randomisation and is expected to be for the duration of the trial:

1. neuroleptics listed in the protocol
2. benzodiazepines and sedatives listed in the protocol

   * Clinically significant uncompensated hearing loss in the judgment of the investigator. Use of hearing aids is allowed.
   * Known hypersensitivity to the drug product excipients

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (52):
- United States (7):
  - Orange County Neuropsychiatric Research Center LLC, Orange, California
  - California Neuroscience Research, Sherman Oaks, California
  - Premiere Research Institute, West Palm Beach, Florida
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Richmond Behavioral Associates, Staten Island, New York
  - ANI Neurology, PLLC, dba Alzheimer's Memory Center, Charlotte, North Carolina
  - Tulsa Clinical Research, LLC, Tulsa, Oklahoma
- Austria (2):
  - Landeskrankenhaus Hall, Abt.f. Psychatrie & Psychotherapie A, Hall in Tirol
  - Private Practice for Psychiatry and Neurology, Vienna
- Brussels-UNIV Brugmann -Horta, Brussels, Belgium
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - Royal Jubilee Hospital, Victoria, British Columbia
  - True North Clinical Research Halifax, Inc., Halifax, Nova Scotia
  - True North Clinical Research Kentville, Inc., Kentville, Nova Scotia
  - Toronto Memory Program, Toronto, Ontario
  - Institut universitaire de geriatrie Sherbrooke, Québec
- France (5):
  - HOP Pierre Wertheimer, Bron
  - HOP Gui de Chauliac, Montpellier
  - HOP Nord Laënnec, Nantes
  - HOP La Pitié Salpêtrière, Paris
  - HOP Jean Bernard, Géria, Poitiers, Poitiers
- Germany (6):
  - Praxis Dr. med. Volker Schumann, Berlin
  - emovis GmbH, Berlin
  - AFL Arzneimittelforschung Leipzig GmbH, Leipzig
  - Zentralinstitut für seelische Gesundheit, Mannheim
  - Universitätsklinikum Ulm, Ulm
  - Neurologie und Psychiatrie / Psychotherapie, Westerstede
- Italy (3):
  - A.O. Spedali Civili di Brescia, Brescia
  - Osp. S. Giovanni di Dio, Florence
  - Policlinico Gemelli, Roma
- Brain Research Center, Amsterdam, Netherlands
- Poland (8):
  - Podlassian Center of Psychogeriatry, Bialystok, Bialystok
  - Non-Public Outpat. Clinic "Dom Sue Ryder", PALLMED Sp. z o.o, Bydgoszcz
  - Non-Public Outpatient Clinic "Synapsa" Pawel Polrola, Kielce, Kielce
  - Mental Health Center Biomed, Kielce
  - Non-Public Outpatient Clinic Neuro-Kard Ilkowski & Partners, Poznan
  - Medical Center Senior, Sopot
  - EUROMEDIS Sp. z o.o., Szczecin, Szczecin
  - Reg. Specialist Hospital Wroclaw, Research & Develop. Center, Wroclaw
- Portugal (4):
  - Hospital Fernando Fonseca, EPE, Amadora
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - CHLO, EPE - Hospital Egas Moniz, Lisbon
  - CHLN, EPE - Hospital de Santa Maria, Lisbon
- Spain (6):
  - Hospital Universitario Fundación Alcorcón, Alcorcon (Madrid)
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Virgen de la Arrixaca, El Palmar (murcia)
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès
  - Hospital Mútua Terrassa, Terrasa (Barcelona)
- United Kingdom (3):
  - Royal United Hospital, Bath
  - Derriford Hospital, Plymouth
  - Re-Cognition Health, Plymouth

REFERENCES:
- [Derived] Frolich L, Wunderlich G, Thamer C, Roehrle M, Garcia M Jr, Dubois B. Evaluation of the efficacy, safety and tolerability of orally administered BI 409306, a novel phosphodiesterase type 9 inhibitor, in two randomised controlled phase II studies in patients with prodromal and mild Alzheimer's disease. Alzheimers Res Ther. 2019 Feb 12;11(1):18. doi: 10.1186/s13195-019-0467-2. PMID 30755255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multi-centre, double-blind, parallel-group, randomized controlled study to investigate the efficacy, safety and tolerability of orally administered BI 409306 during a 12-week treatment period compared to placebo in patients with Alzheimer's Disease
Pre-assignment Details: For this trial, patients were randomised at 36 sites in 11 countries. Following an initial Screening Visit and a single blinded 2-week placebo run-in period, patients who qualified according to the in- and exclusion criteria were randomised to one of the five treatment groups
Groups:
- BI 409306 10 Milligram (mg) Once Daily (QD): Patients were administered orally a tablet of 10 mg BI 409306 once daily for 12 weeks.
- BI 409306 25 mg QD: Patients were administered orally a tablet of 25 mg BI 409306 once daily for 12 weeks.
- BI 409306 50 mg QD: Patients were administered orally a tablet of 50 mg BI 409306 once daily for 12 weeks.
- BI 409306 25 mg Twice Daily (BID): Patients were administered orally a tablet of 25 mg BI 409306 twice daily for 12 weeks.
- Placebo Matching BI 409306: Patients were administered orally Placebo matching 10 mg/25 mg/ 50 mg BI 409306 for 12 weeks
Period: Overall Study
Arm/Group | BI 409306 10 Milligram (mg) Once Daily (QD) | BI 409306 25 mg QD | BI 409306 50 mg QD | BI 409306 25 mg Twice Daily (BID) | Placebo Matching BI 409306
Started | 22 | 21 | 21 | 21 | 43
Completed | 22 | 21 | 17 | 20 | 42
Not Completed | 0 | 0 | 4 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1 | 0
Not completed — Other than specified | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set:
  The treated set (TS) included all patients who were randomised and treated with at least one dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 409306 10 Milligram (mg) Once Daily (QD) | BI 409306 25 mg QD | BI 409306 50 mg QD | BI 409306 25 mg Twice Daily (BID) | Placebo Matching BI 409306 | Total
Number analyzed (Participants) | 22 | 21 | 21 | 21 | 43 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.3 (5.4) | 74.1 (8.1) | 73.3 (5.1) | 71.9 (6.0) | 72.2 (6.5) | 72.7 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 8 | 13 | 28 | 71
  Male | 12 | 9 | 13 | 8 | 15 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race data is presented below; Ethnicity was not reported in this trial
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0
    White | 22 | 21 | 21 | 21 | 43 | 128
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Neuropsychological Test Battery (NTB) Total [Mean (Standard Deviation); unit: z-score] — Baseline cognitive assessment data- NTB total z-score. The NTB consists of 9 validated components. Raw scores on each of the 9 NTB tests were converted to z-scores using the baseline means and standard deviations (SDs) for each test. The resultant z-scores were averaged to obtain a total z-score, incorporating all 9 NTB tests. The NTB Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean at baseline. Higher values indicate a better Outcome
  z-score | 0.07 (0.70) | 0.02 (0.75) | -0.02 (0.72) | -0.02 (0.61) | -0.03 (0.63) | -0.00 (0.66)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Neuropsychological Test Battery in Total Z-score After 12-week Treatment.
Description: Neuropsychological Test Battery (NTB) response, defined as change from baseline in total z-score after 12 weeks of treatment. The NTB Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean at baseline. Negative numbers indicate values lower than baseline and positive numbers indicate values higher than baseline. Change from baseline will be calculated as the post-baseline composite z-score minus the pre-treatment z-score, such that a positive change indicates an improvement from baseline
Time Frame: Baseline and 12 weeks
Population: The full analysis set (FAS) included all randomised patients who were treated with at least one dose of trial medication and had a baseline and at least one post-baseline on-treatment efficacy assessment. Observed cases (OC)
Measure: Least Squares Mean (Standard Error); unit: z-score
Groups:
- Pooled BI 409306: Patients were administered orally a tablet of BI 409306 (10 mg, 25 mg, 50 mg once daily and 25 mg twice daily)for 12 weeks.
Arm/Group | BI 409306 10 Milligram (mg) Once Daily (QD) | BI 409306 25 mg QD | BI 409306 50 mg QD | BI 409306 25 mg Twice Daily (BID) | Pooled BI 409306 | Placebo Matching BI 409306
Number analyzed (Participants) | 20 | 19 | 16 | 18 | 73 | 39
z-score | 0.35 (0.061) | 0.20 (0.063) | 0.26 (0.065) | 0.32 (0.064) | 0.29 (0.031) | 0.27 (0.043)
Statistical Analysis 1: Comparison: BI 409306 10 Milligram (mg) Once Daily (QD) vs Placebo Matching BI 409306; Mixed Model Repeated Measurement (MMRM) includes fixed, categorical effects of treatment, visit, and treatment-by-visit interaction, as well as the continuous fixed covariates of baseline, and baseline-by-visit interaction; Test type: Superiority — H0: The dose group with the peak response in the respective model Mean NTB response = Mean NTB response of placebo; p = 0.3236, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.074 to 0.223], Standard Error of Mean 0.075 — Mean difference (BI 409306 10 milligram (mg) once daily (QD) minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 2: Comparison: BI 409306 25 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — H0: The dose group with the peak response in the respective model Mean NTB response = Mean NTB response of placebo; p = 0.3694, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.220 to 0.082], Standard Error of Mean 0.076 — Mean difference (BI 409306 25 mg QD minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 3: Comparison: BI 409306 50 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — H0: The dose group with the peak response in the respective model Mean NTB response = Mean NTB response of placebo; p = 0.8374, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.171 to 0.139], Standard Error of Mean 0.078 — Mean difference (BI 409306 50 mg QD minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 4: Comparison: BI 409306 25 mg Twice Daily (BID) vs Placebo Matching BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — H0: The dose group with the peak response in the respective model Mean NTB response = Mean NTB response of placebo; p = 0.5484, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.106 to 0.199], Standard Error of Mean 0.077 — Mean difference (BI 409306 25 mg twice daily (BID) minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 5: Comparison: Pooled BI 409306 vs Placebo Matching BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — H0: The dose group with the peak response in the respective model Mean NTB response = Mean NTB response of placebo; p = 0.7905, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.092 to 0.121], Standard Error of Mean 0.054 — Mean difference (Pooled BI 409306 minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences

2. Secondary Outcome: Change From Baseline in ADCS-MCI-ADL (Alzheimer's Disease Cooperative Study/Activities of Daily Living for Patients With Mild Cognitive Impairment) Total Score After 12-week Treatment
Description: Alzheimer's Disease Cooperative Study/Activities of Daily Living (ADCS-ADL) is a rating scale used to assess basic and instrumental activities of daily living. In the full version of the scale, 23 items are rated by the investigator using information supplied by the caregiver.
  Each item has a score range varying from 0-3 to 0-5. The sum score can range from 0 to 78. Higher scores indicate better function.
  Least Squares Mean is actually an adjusted mean change from baseline.
Time Frame: Baseline and 12 weeks
Population: FAS- Observed cases
Measure: Least Squares Mean (Standard Error); unit: Unit on scale
Arm/Group | BI 409306 10 Milligram (mg) Once Daily (QD) | BI 409306 25 mg QD | BI 409306 50 mg QD | BI 409306 25 mg Twice Daily (BID) | Placebo Matching BI 409306
Number analyzed (Participants) | 19 | 18 | 20 | 17 | 37
Unit on scale | 0.24 (0.896) | 1.79 (0.921) | -0.10 (0.875) | 0.80 (0.947) | 0.38 (0.642)
Statistical Analysis 1: Comparison: BI 409306 10 Milligram (mg) Once Daily (QD) vs Placebo Matching BI 409306; The dependent variable was the change from the baseline score at Week 12. The model included fixed, categorical covariates of treatment as well as fixed continuous covariates of baseline score; Test type: Superiority — Analyses of covariance (ANCOVA) were used to assess between-group differences in the modelled changes from baseline to Week 12; p = 0.8973, ANCOVA — p-value was nominal and not adjusted; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-2.33 to 2.04], Standard Error of Mean 1.102 — Mean difference (BI 409306 10 milligram (mg) once daily (QD) minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 2: Comparison: BI 409306 25 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.2141, ANCOVA — p-value was nominal and not adjusted; Mean Difference (Final Values) = 1.40, 95% CI 2-sided [-0.82 to 3.63], Standard Error of Mean 1.122 — Mean difference (BI 409306 25 mg QD minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 3: Comparison: BI 409306 50 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.6553, ANCOVA — p-value was nominal and not adjusted; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-2.64 to 1.67], Standard Error of Mean 1.085 — Mean difference (BI 409306 50 mg QD minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 4: Comparison: BI 409306 25 mg Twice Daily (BID) vs Placebo Matching BI 409306; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.7166, ANCOVA — p-value was nominal and not adjusted; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-1.85 to 2.69], Standard Error of Mean 1.144 — Mean difference (BI 409306 25 mg twice daily (BID) minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences

3. Secondary Outcome: Change From Baseline in Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) Total Score After 12-week Treatment
Description: The CDR-SB is obtained through semi-structured interviews of patients and informants, and cognitive functioning was rated in 6 domains of functioning: memory, orientation, judgment and problem solving, community affairs, home and hobbies and personal care.
  Each domain was rated on a 5-point scale of functioning as follows: 0-no impairment; 0.5-questionable impairment; 1-mild impairment; 2-moderate impairment and 3-severe impairment. Only personal care was scored on a 4-point scale without a 0.5 rating available. The higher the score, the greater the severity of dementia. Least Squares Mean is actually an adjusted mean change from baseline.
Time Frame: Baseline and 12 weeks
Population: FAS- Observed cases
Measure: Least Squares Mean (Standard Error); unit: Unit on scale
Arm/Group | BI 409306 10 Milligram (mg) Once Daily (QD) | BI 409306 25 mg QD | BI 409306 50 mg QD | BI 409306 25 mg Twice Daily (BID) | Placebo Matching BI 409306
Number analyzed (Participants) | 21 | 19 | 16 | 18 | 40
Unit on scale | 0.0 (0.19) | 0.4 (0.20) | -0.1 (0.22) | 0.1 (0.21) | 0.1 (0.14)
Statistical Analysis 1: Comparison: BI 409306 10 Milligram (mg) Once Daily (QD) vs Placebo Matching BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.9491, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.49 to 0.46], Standard Error of Mean 0.24 — Mean difference (BI 409306 10 milligram (mg) once daily (QD) minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 2: Comparison: BI 409306 25 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1699, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.15 to 0.84], Standard Error of Mean 0.25 — Mean difference (BI 409306 25 mg QD minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 3: Comparison: BI 409306 50 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4948, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.69 to 0.33], Standard Error of Mean 0.26 — Mean difference (BI 409306 50 mg QD minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 4: Comparison: BI 409306 25 mg Twice Daily (BID) vs Placebo Matching BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.7548, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.42 to 0.58], Standard Error of Mean 0.25 — Mean difference (BI 409306 25 mg twice daily (BID) minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences

4. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-cognitive Subscale (ADAS-cog11) Total Score After 12-week Treatment
Description: Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog11) is an 11-item cognitive subscale that objectively measures memory, language, orientation, and praxis with a total score range of 0 to 70. The greater the dysfunction, the greater the score. Least Squares Mean is actually an adjusted mean change from baseline.
Time Frame: Baseline and 12 weeks
Population: FAS- Observed cases
Measure: Least Squares Mean (Standard Error); unit: Unit on scale
Arm/Group | BI 409306 10 Milligram (mg) Once Daily (QD) | BI 409306 25 mg QD | BI 409306 50 mg QD | BI 409306 25 mg Twice Daily (BID) | Placebo Matching BI 409306
Number analyzed (Participants) | 19 | 17 | 19 | 19 | 38
Unit on scale | 0.98 (0.885) | 0.62 (0.935) | 0.12 (0.875) | -1.27 (0.875) | 1.24 (0.619)
Statistical Analysis 1: Comparison: BI 409306 10 Milligram (mg) Once Daily (QD) vs Placebo Matching BI 409306; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.8137, ANCOVA — p-value was nominal and not adjusted; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-2.40 to 1.89], Standard Error of Mean 1.081 — Mean difference (BI 409306 10 milligram (mg) once daily (QD) minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 2: Comparison: BI 409306 25 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.5801, ANCOVA — p-value was nominal and not adjusted; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-2.84 to 1.60], Standard Error of Mean 1.120 — Mean difference (BI 409306 25 mg QD minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 3: Comparison: BI 409306 50 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.2978, ANCOVA — p-value was nominal and not adjusted; Mean Difference (Final Values) = -1.12, 95% CI 2-sided [-3.25 to 1.00], Standard Error of Mean 1.072 — Mean difference (BI 409306 50 mg QD minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 4: Comparison: BI 409306 25 mg Twice Daily (BID) vs Placebo Matching BI 409306; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0209, ANCOVA — p-value was nominal and not adjusted; Mean Difference (Final Values) = -2.51, 95% CI 2-sided [-4.64 to -0.39], Standard Error of Mean 1.072 — Mean difference (BI 409306 25 mg twice daily (BID) minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences

5. Primary Outcome: Change From Baseline in Neuropsychological Test Battery in Total Z-score After 12-week Treatment From Two Twin Trials, Present 1289.5 (NCT02240693) and 1289.7 (NCT02337907)
Description: as for outcome 1
Time Frame: Baseline and 12 weeks
Population: FAS observed cases for pooled groups of these twin trials
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | BI 409306 10 Milligram (mg) Once Daily (QD) | BI 409306 25 mg QD | BI 409306 50 mg QD | BI 409306 25 mg Twice Daily (BID) | Pooled BI 409306 | Placebo Matching BI 409306
Number analyzed (Participants) | 67 | 63 | 67 | 63 | 260 | 122
z-score | 0.20 (0.046) | 0.19 (0.048) | 0.19 (0.046) | 0.10 (0.047) | 0.17 (0.025) | 0.19 (0.035)
Statistical Analysis 1: Comparison: BI 409306 10 Milligram (mg) Once Daily (QD) vs Placebo Matching BI 409306; Mixed Model Repeated Measurement (MMRM) includes fixed, categorical effects of treatment, visit, current Acetylcholine Esterase Inhibitor (AChEI) use (Yes, No), and treatment-by-visit interaction, as well as the continuous fixed covariates of baseline, and baseline-by-visit interaction. The study identifier is also a categorical covariate for the twin studies analyses; Test type: Superiority — H0: The dose group with the peak response in the respective model Mean NTB response = Mean NTB response of placebo; p = 0.8694, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.101 to 0.120], Standard Error of Mean 0.056 — Mean difference (BI 409306 10 milligram (mg) once daily (QD) minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 2: Comparison: BI 409306 25 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 5, analysis 1]; Test type: Superiority — H0: The dose group with the peak response in the respective model Mean NTB response = Mean NTB response of placebo; p = 0.9512, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.116 to 0.109], Standard Error of Mean 0.057 — Mean difference (BI 409306 25 mg QD minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 3: Comparison: BI 409306 50 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 5, analysis 1]; Test type: Superiority — H0: The dose group with the peak response in the respective model Mean NTB response = Mean NTB response of placebo; p = 0.9321, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.105 to 0.115], Standard Error of Mean 0.056 — Mean difference (BI 409306 50 mg QD minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 4: Comparison: BI 409306 25 mg Twice Daily (BID) vs Placebo Matching BI 409306; [analysis description as in outcome 5, analysis 1]; Test type: Superiority — H0: The dose group with the peak response in the respective model Mean NTB response = Mean NTB response of placebo; p = 0.1288, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.199 to 0.025], Standard Error of Mean 0.057 — Mean difference (BI 409306 25 mg twice daily (BID) minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 5: Comparison: Pooled BI 409306 vs Placebo Matching BI 409306; [analysis description as in outcome 5, analysis 1]; Test type: Superiority — H0: The dose group with the peak response in the respective model Mean NTB response = Mean NTB response of placebo; p = 0.6492, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.098 to 0.061], Standard Error of Mean 0.041 — Mean difference (Pooled BI 409306 minus Placebo matching BI 409306); The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences

ADVERSE EVENTS:
Time Frame: From the first dose of study medication until 7 days after last administration of BI 409306, up to 16 weeks.
Description: The treated set (TS) used (all patients who were randomised and treated with at least one dose of trial medication.) for safety assessment.
Groups:
- Placebo Matching BI 409306: Patients were administered orally tablet of Placebo matching BI 409306 once daily for 12 weeks.
Arm/Group | BI 409306 10 Milligram (mg) Once Daily (QD) | BI 409306 25 mg QD | BI 409306 50 mg QD | BI 409306 25 mg Twice Daily (BID) | Placebo Matching BI 409306
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/21 | 0/21 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/21 | 1/21 | 1/43
Other Adverse Events (participants affected / at risk) | 5/22 | 8/21 | 11/21 | 3/21 | 6/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 409306 10 Milligram (mg) Once Daily (QD) (N=22) | BI 409306 25 mg QD (N=21) | BI 409306 50 mg QD (N=21) | BI 409306 25 mg Twice Daily (BID) (N=21) | Placebo Matching BI 409306 (N=43)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 409306 10 Milligram (mg) Once Daily (QD) (N=22) | BI 409306 25 mg QD (N=21) | BI 409306 50 mg QD (N=21) | BI 409306 25 mg Twice Daily (BID) (N=21) | Placebo Matching BI 409306 (N=43)
Bradycardia (Cardiac disorders) | 2 | 3 | 1 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 4 | 3 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 2 | 0 | 4 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT02240693/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT02240693/SAP_001.pdf